CLINICAL TRIAL: NCT05064072
Title: The Evaluation of Pain Felt During Removal of the Products From Infant's Skin Used in Nasogastric Tube Fixation: Randomized Controlled Study
Brief Title: Pain Felt During Removal of the Products From Infant's Skin Used in Nasogastric Tube Fixation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23618724
Record Dates: First submitted 2021-09-29; First posted 2021-10-01 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Pain, Acute
Keywords: infant; pain; adhesives; fixation
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Water-based barrier tape (Experimental): The infants in experiment 1 group will be applied water-based barrier tape will be used to fix the nasogastric tube
  Interventions: Device: Water-based barrier tape
- Hydrocolloid barrier tape (Experimental): The infants in experiment 2 group, hydrocolloid barrier tape will be used to fix the nasogastric tube
  Interventions: Device: Hydrocolloid barrier tape
- Silk plaster (Active Comparator): The silk plaster used in clinic routinely will be used for control group infants to fix the nasogastric tube
  Interventions: Device: Silk tape

INTERVENTIONS:
Device: Water-based barrier tape — The infants in experiment 1 group will be applied water-based barrier tape. The area will be covered by water-based barrier tape to fix nasogastric tube and after waiting 1 minute for drying up it will be fastened by silk tape used in clinic. The silk tape will be 5 cm long and it will be changed in every 24 hours. Following the removal of silk tape on the water-based barrier tape, the pain felt by the infants evaluated through "Neonatal Infant Pain Scale" and the score recorded in the chart. This procedure actualized 3 min. before procedure, during and 3 min after procedure.
  Arms: Water-based barrier tape
Device: Hydrocolloid barrier tape — As for experiment 2 group, hydrocolloid barrier tape will be used to fix the nasogastric tube. The hydrocolloid barrier tape, which was cut and shaped appropriately beforehand, will be applied to the area in order to stabilize the nasogastric tube and the tube will be stabilized with silk tape used in clinic. The silk tape will be 5 cm long and it will be changed in every 24 hours. Following the removal of silk tape on the hydrocolloid barrier tape, the pain felt by the infants evaluated with "Neonatal Infant Pain Scale" and the score recorded in the chart. Since the hydrocolloid barrier tape can stay on the skin for 7 days and the assessment of the pain realized in 7th day and noted down to the chart. Pain score evaluated in 7th day 3 min. before procedure, during and 3 min after procedure
  Arms: Hydrocolloid barrier tape
Device: Silk tape — The silk tape used in clinic routinely will be used for control group infants to fix the nasogastric tube without any barrier. The silk tape will be 5cm long and it will be changed in every 24 hours. Following the removal of silk tape on the silk tape, the pain felt by the infants evaluated through "Neonatal Infant Pain Scale" and the score recorded in the chart. This procedure actualized 3 min. before procedure, during and 3 min after procedure
  Arms: Silk plaster

SUMMARY:
The present study was planned to evaluate the pain of 4-6 weeks infants felt during removal of the adhesive products from newborn's skin used in the fixation of nasogastric tube in neonatal and infant units. The hypothesis of the study is "Water-based barrier tape is more effective to reduce pain than hydrocolloid barrier tape.

DETAILED DESCRIPTION:
The study was planned as randomized controlled and experimental design to compare the efficiency of three different methods reducing pain during removal adhesive products for 4-6 weeks infants. The universe of the study consisted of 4-6 weeks infants in neonatal and infants clinics of Giresun Women's and Children's Hospital between the dates of July-September 2021. Power analysis was performed through G*Power (v3.1.7) programme in order to determine the number of the sample. At the beginning of the study, a reference study (Kemer, 2020) was used for sample calculation. The effect size was calculated as d=0.561 regarding the assessment of skin condition scores and 120 participants in total should be included in the study as 40 participants for each groups in order to obtain 80% power in the level of α=0.05. Block randomization technique is applied in the study as a randomization method. "As for data collection "Infant description form" and "Neonatal Infant Pain Scale" was used. The scale was filled by two independent observer via double-blind method.

ELIGIBILITY:
Inclusion Criteria:

* All the 4-6 weeks infants including interventional process and without any skin diseases

Exclusion Criteria:

* The infants receiving treatment without any interventional process
* Those having a skin disease
* Those infants having peripherally inserted central venous catheter

Ages: 4 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Water-based barrier tape | 24 hours
  To evaluate pain felt by infants following the removal of silk adhesive from water-based barrier tape
Hydrocolloid barrier tape | 24 hours
  To evaluate pain felt by infants following the removal of silk adhesive from hydrocolloid barrier tape
Silk Tape | 24 hours
  To evaluate pain felt by infants following the removal of silk adhesive from infants skin without any barrier tape

CONTACTS AND LOCATIONS:
Locations (1):
- Giresun University Women and Children's Hospital, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Field T. Preterm newborn pain research review. Infant Behav Dev. 2017 Nov;49:141-150. doi: 10.1016/j.infbeh.2017.09.002. Epub 2017 Sep 9. PMID 28898671
- [Result] Maxwell LG, Fraga MV, Malavolta CP. Assessment of Pain in the Newborn: An Update. Clin Perinatol. 2019 Dec;46(4):693-707. doi: 10.1016/j.clp.2019.08.005. Epub 2019 Aug 19. PMID 31653303
- [Result] Kemer D, İşler Dalgıç A. Yenidoğanlarda Ağrı Yönetiminde Kullanılan Kanıt Temelli Non-Farmakolojik Hemşirelik Uygulamaları. Balıkesir Sağlık Bilimleri Dergisi. 2020; 9(3):197-204.